CLINICAL TRIAL: NCT04571528
Title: Effectiveness of Virtual Multicomponent Treatment for Fibromyalgia: VIRTUAL FIBROWALK STUDY
Brief Title: Effectiveness of VIRTUAL FIBROWALK STUDY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PR(AG)249/2020
Record Dates: First submitted 2020-09-25; First posted 2020-10-01 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Fibromyalgia
Keywords: multicomponent treatment; Fibromyalgia; chronic pain; pain neuroscience education; therapeutic exercise; cognitive behavioural therapy; mindfulness; randomized controlled trial
MeSH Terms: conditions — Fibromyalgia; Chronic Pain | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Parallel Assignment Single-blind, parallel-group, randomized controlled trial
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TAU + multicomponent treatment VIRTUAL FIBROWALK (Experimental): VIRTUAL FIBROWALK is a multicomponent non-pharmacological program based on Pain Neuroscience Education (PNE), therapeutic exercise, Cognitive Behavioural Therapy (CBT) and Mindfulness Training
  Interventions: Behavioral: TAU + multicomponent treatment VIRTUAL FIBROWALK
- Treatment as Usual (TAU) (Active Comparator): Treatment-as-Usual (TAU) consisted of the prescribed drugs adapted to the symptomatic profile of each patient and basic face to face and written advice on PNE and aerobic exercise adapted to the physical capacities of the patients at the beginning of the study.patient
  Interventions: Behavioral: Treatment as Usual (TAU)
- Physiotherapy part of VIRTUA FIBROWALK (Active Comparator): The physiotherapy part of the VIRTUAL FIBROWALK is a multicomponent non-pharmacological program based on Pain Neuroscience Education (PNE) and therapeutic exercise.
  Interventions: Behavioral: TAU + Physiotherapy part of VIRTUAL FIBROWALK

INTERVENTIONS:
Behavioral: TAU + multicomponent treatment VIRTUAL FIBROWALK — Group treatment protocol of 12 weekly 60 minute virtual sessions. All sessions include the following ingredients (approx. in the same order): - Pain neuroscience education (15 min.) - Cognitive restructuring (15 min.) - Mindfulness techniques (15 min.) - Physical exercise(15 min.) - Treatment as Usual (TAU) Standard pharmacological treatment usually provided to patients with fibromyalgia.
  Arms: TAU + multicomponent treatment VIRTUAL FIBROWALK
Behavioral: Treatment as Usual (TAU) — Treatment-as-Usual (TAU) consisted of the prescribed drugs adapted to the symptomatic profile of each patient and basic face to face and written advice on PNE and aerobic exercise adapted to the physical capacities of the patients at the beginning of the study.
  Arms: Treatment as Usual (TAU)
Behavioral: TAU + Physiotherapy part of VIRTUAL FIBROWALK — Group treatment protocol of 12 weekly 60 minute virtual sessions. All sessions include the following ingredients: - Pain neuroscience education (30 min.) - Physical exercise(30 min.) - Treatment as Usual (TAU). Standard pharmacological treatment usually provided to patients with fibromyalgia.
  Arms: Physiotherapy part of VIRTUA FIBROWALK

SUMMARY:
The main objective of this study is to analyse the effectiveness of the VIRTUAL FIBROWALK multicomponent treatment program as coadjuvant of treatment-as-usual (TAU) compared to TAU alone. In this Randomized Controlled Trial (RCT), in addition to evaluating the clinical effects of VIRTUAL FIBROWALK treatment in the short- and longterm.

DETAILED DESCRIPTION:
This is a tree-arm RCT focused on the safety and potential effectiveness of the multicomponent program VIRTUAL FIBROWALK as coadjuvant of treatment-as-usual (TAU) vs. TAU alone and on the comparation of the physiotherapy part of the multicomponent program.

* VIRTUAL FIBROWALK combines multicomponent approach based on Pain Neuroscience Education (PNE), therapeutic exercise, Cognitive Behavioural Therapy (CBT) and Mindfulness training.
* Physiotherapy part of VIRTUAL FIBROWALK combines multicomponent approach based on Pain Neuroscience Education (PNE) and therapeutic exercise.
* The main hypothesis is that improvement on functional impairment of patients with fibromyalgia can be achieved by the direct intervention on mechanisms such as kinesiophobia and fear avoidance

ELIGIBILITY:
Inclusion Criteria:

* Adults from 18 to 75 years-old.
* 1990 American College of Rheumatology (ACR) classification criteria + the 2011 modified ACR diagnostic criteria for fibromyalgia
* Able to understand Spanish and accept to participate in the study.

Exclusion Criteria:

* Participating in concurrent or past RCTs (previous year).
* Comorbidity with severe mental disorders (i.e. psychosis) or neurodegenerative diseases (i.e. Alzheimer) that that would limit the ability of the patient to participate in the RCT.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-09-21 (Actual); Primary Completion 2021-11-10 (Estimated); Study Completion 2021-11-10 (Estimated)

PRIMARY OUTCOMES:
Revised Fibromyalgia Impact Questionnaire (FIQR) | Through study completion, an average of 3 months
  The FIQR comprises three dimensions: physical dysfunction (scores from 0 to 30), overall impact (scores from 0 to 20), and intensity of the symptoms (scores from 0 to 50) is used to measure the impact generated by FM during the last week. It consists of 21 items, which are answered on a numerical rating scale of 11 points (from 0 to 10). Total scores can range from 0 to 100, with higher scores reflecting greater deterioration.

SECONDARY OUTCOMES:
Tampa Scale for Kinesiophobia (TSK-11) | Through study completion, an average of 3 months
  TSK-11 is used to assess fear of pain and movement. It consists of 11 items, which are answered on a Likert scale of 4 points. Total scores of each scale range from 11 to 44, where higher scores indicate a greater fear of pain and movement.
Hospital Anxiety and Depression Scale (HADS) | Through study completion, an average of 3 months
  HADS is used to quantify the severity of anxiety and depression symptoms. It consists of two dimensions (anxiety and depression) of 7 items each responding on a Likert scale of 4 points. Total scores of each scale (HADS-A and HADSD) range from 0 to 21, where higher scores indicate greater severity of symptoms.
Physical Function of the 36-Item Short Form Survey (SF-36) | Through study completion, an average of 3 months
  Physical Function of the 36-Item Short Form Survey (SF-36) was used to measure physical function.This dimension comprises a total of 10 items, which are answered on a Likert scale of 3 points. Total scores on each scale are then transformed and can range from 0 to 100, with higher scores indicate better physical function.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Marsal, PhD, Principal Investigator — Vall d'Hebrón Hospital
Locations (1):
- Vall d'Hebrón Hospital, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Serrat M, Albajes K, Navarrete J, Almirall M, Lluch Girbes E, Neblett R, Luciano JV, Moix J, Feliu-Soler A. Effectiveness of two video-based multicomponent treatments for fibromyalgia: The added value of cognitive restructuring and mindfulness in a three-arm randomised controlled trial. Behav Res Ther. 2022 Nov;158:104188. doi: 10.1016/j.brat.2022.104188. Epub 2022 Sep 8. PMID 36116229